CLINICAL TRIAL: NCT00294203
Title: Placebo-Controlled Pilot Study to Assess the Post-Operative Administration of Epoetin Alfa on Patients Undergoing Abdominal or Pelvic Surgery for Malignancy
Brief Title: Pilot Study of Epoetin Alfa for Patients Having Abdominal or Pelvic Surgery for Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPOSUR; 20052318
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Anemia
Keywords: Digestive System Surgical Procedures; Post-Operative Care; Fatigue; Quality of Life; Erythrocyte Transfusion; Esophagectomy; Gastric Cancer; Hepatectomy; Pancreatic Cancer; Rectum
MeSH Terms: conditions — Anemia; Fatigue; Stomach Neoplasms; Pancreatic Neoplasms | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epoetin Alfa group (Active Comparator): Patients enrolled in the study will be randomized to receive either 40,000 units of epoetin alfa on day 1 and day 8. Hemoglobin, hematocrit, reticulocyte count, reticulocyte hemoglobin, and immature reticulocyte count will be measured on days 1, 4, 8, and once between post-operative days 20 and 30. Pre-operatively and between post-operative days 20 and 30 patients will complete a quality of live assessment tool (FACT-An) to assess their fatigue related to anemia.
  Interventions: Drug: Epoetin Alfa group
- Placebo group (Placebo Comparator): Patients enrolled in the study will be randomized to receive either 40,000 units of placebo (saline) on day 1 and day 8. Hemoglobin, hematocrit, reticulocyte count, reticulocyte hemoglobin, and immature reticulocyte count will be measured on days 1, 4, 8, and once between post-operative days 20 and 30. Pre-operatively and between post-operative days 20 and 30 patients will complete a quality of live assessment tool (FACT-An) to assess their fatigue related to anemia.
  Interventions: Other: Placebo group

INTERVENTIONS:
Drug: Epoetin Alfa group — Patients enrolled in the study will be randomized to receive either 40,000 units of epoetin alfa on day 1 and day 8. Hemoglobin, hematocrit, reticulocyte count, reticulocyte hemoglobin, and immature reticulocyte count will be measured on days 1, 4, 8, and once between post-operative days 20 and 30. Pre-operatively and between post-operative days 20 and 30 patients will complete a quality of live assessment tool (FACT-An) to assess their fatigue related to anemia.
  Arms: Epoetin Alfa group
Other: Placebo group — Patients enrolled in the study will be randomized to receive either 40,000 units of placebo (saline) on day 1 and day 8. Hemoglobin, hematocrit, reticulocyte count, reticulocyte hemoglobin, and immature reticulocyte count will be measured on days 1, 4, 8, and once between post-operative days 20 and 30. Pre-operatively and between post-operative days 20 and 30 patients will complete a quality of live assessment tool (FACT-An) to assess their fatigue related to anemia.
  Other Names: saline
  Arms: Placebo group

SUMMARY:
This pilot study is looking at how well epoetin alfa, given in the immediate post-operative period, works in reducing anemia and the need for transfusions.

DETAILED DESCRIPTION:
This is a pilot, single center, prospective, double blinded, randomized study comparing epoetin alfa versus placebo. Eligible patients will just have undergone a major abdominal operation for malignancy (esophagectomy, gastrectomy, partial hepatectomy, partial pancreatectomy, or low anterior resection of rectum) and have a post-operative hemoglobin greater than 8 g/dL and less than 11 g/dL on post-operative day #1. On post-operative day #1 patients enrolled in the study will be randomized to receive either 40,000 units of epoetin alfa or placebo. On post-operative day #8, the patients will receive an additional dose of epoetin alfa or placebo (depending on randomization assignment and Hgb level). Hemoglobin, hematocrit, reticulocyte count, reticulocyte hemoglobin, and immature reticulocyte count will be measured on days 1, 4, 8, and once between post-operative days 20 and 30. Pre-operatively and between post-operative days 20 and 30 patients will complete a quality of live assessment tool (FACT-An) to assess their fatigue related to anemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing esophagectomy, gastrectomy, partial pancreatectomy, hepatic resection, or low anterior resection of rectum for malignancy
* Patients with hemoglobin greater than 8 and less than 11 g/dL on post-operative day #1.

Exclusion Criteria:

* Patients receiving red blood cell transfusion within the first twelve hours post-operatively.
* Patients receiving epoetin-stimulating proteins within 30 days prior to the operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Post-operative hemoglobin, reticulocyte count, reticulocyte hemoglobin, and immature reticulocyte fraction measured on post-operative days 1, 4, 8, and between days 20 and 30 | 1,4,8 and between 20 and 30 days post op

SECONDARY OUTCOMES:
Post-operative quality of life related to anemia measured by Functional Assessment of Cancer Therapy - Anemia (FACT-An) between post-operative day 20 and 30 and post-operative transfusion requirement | between 20 and 30 days postop

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R. Grobmyer, MD, Principal Investigator — University of Florida Division of Surgical Oncology and Endocrine Surgery
Locations (2):
- United States (2):
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida